CLINICAL TRIAL: NCT01053715
Title: A European, Prospective, Non-Interventional Study to Assess Health Related Quality of Life and to Identify Key Transitional Life Events in Patients With Moderate or Severe Haemophilia A Using Helixate NexGen
Brief Title: Quality of Life Study of Helixate NexGen
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CE1250_5002_EU; 1501 (Other: CSL Behring)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Hemophilia A
Keywords: Hemophilia; Quality of Life
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe Health Related Quality of Life (HRQoL) in adolescents and adults with Hemophilia A treated prophylactically or on-demand with Helixate NexGen. The study will also assess the kinds of determinants, including key transitional life events, that might impact HRQoL in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A patient
* Severely (<1%) and moderately (1-5%) affected
* On treatment with Helixate NexGen
* Ability to read and understand study materials (patient information and data protection form, patient-related questionnaires)
* Signed data protection form; if patient is <18 years of age, legal guardian must also give written consent by signing the data protection form

Exclusion Criteria:

* Presence of inhibitors
* Abuse of recreational drugs or alcohol interfering with the every-day-life in the opinion of the physician
* Advanced stage human immunodeficiency virus (HIV) infection (CD4 cell counts <200/cmm, multi-drug resistance, presence of AIDS related signs or symptoms)
* Symptomatic liver disease (cirrhosis, ascites, esophageal varices)
* Concomitant or planned interferon therapy
* Malignancies on or off treatment

Ages: 14 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a diagnosis of moderate or severe Hemophilia A using Helixate NexGen identified by selected European hemophilia treatment centers.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQoL) | baseline and every 12 months over 3 years

SECONDARY OUTCOMES:
Change in HRQoL due to pre-specified factors potentially affecting HRQoL in patients with hemophilia | Duration of the study
Change in HRQoL due to transitional life events | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klamroth, MD, Principal Investigator — Hämophiliezentrum, Vivantes-Klinikum im Friedrichshain Zentrum für Gefäßmedizin, Berlin; Alessandro Gringeri, MD, Principal Investigator — I.R.C.C.S. Fondazione Ospedale Maggiore Policlinico, Milan
Locations (31):
- Austria (9):
  - CSLB Study Site 22, Graz
  - CSLB Study Site 26, Grieskirchen
  - CSLB Study Site 24, Innsbruck
  - CSLB Study Site 29, Klagenfurt
  - CSLB Study Site 23, Linz
  - CSLB Study Site 25, Sankt Pölten
  - CSLB Study Site 20, Vienna
  - CSLB Study Site 21, Vienna
  - CSLB Study Site 27, Vienna
- Belgium (2):
  - CSLB Study Site 52, Edegem
  - CSLB Study Site 51, Leuven
- France (5):
  - CSLB Study Site 65, Amiens
  - CSLB Study Site 68, Poitiers
  - CSLB Study Site 60, Rouen
  - CSLB Study Site 64, Strasbourg
  - CSLB Study Site 66, Valence
- Germany (6):
  - CSLB Study Site 1, Berlin
  - CSLB Study Site 3, Bonn
  - CSLB Study Site 2, Bremen
  - CSLB Study Site 6, Delmenhorst
  - CSLB Study Site 7, Göttingen
  - CSLB Study Site 4, München
- Italy (4):
  - CSLB Study Site 72, Genova
  - CSLB Study Site 71, Milan
  - CSLB Study Site 74, Napoli
  - CSLB Study Site 73, Palermo
- Spain (3):
  - CSLB Study Site 98, Badajoz
  - CSLB Study Site 95, Jaén
  - CSLB Study Site 91, Valencia
- Switzerland (2):
  - CSLB Study Site 35, Sankt Gallen
  - CSLB Study Site 36, Zurich